CLINICAL TRIAL: NCT05468931
Title: Prostate Stimulation for Sexual Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Eisenberg, Study Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 65918
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Sexual Dysfunction; Erectile Dysfunction; Delayed Ejaculation; Anorgasmia
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Erectile Dysfunction; Ejaculatory Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate stimulation device arm (Experimental): Participants will be asked to use our prostate stimulation device.
  Interventions: Device: Prostate stimulator

INTERVENTIONS:
Device: Prostate stimulator — Prostate stimulation device for sexual dysfunction

SUMMARY:
The purpose of this study is to use a device to stimulate the prostate with a goal of helping improve symptoms in men with sexual dysfunction.

DETAILED DESCRIPTION:
The purpose of the study is to use a device to stimulate the prostate. The goal of this is to help men with sexual dysfunction. Sexual dysfunction can include conditions like delayed ejaculation (e.g.takes more than 21 minutes to climax) and can hopefully assist them in achieving faster time to ejaculation (e.g. closer to the median of 5.4 minutes in a "normal" individual) along with erectile dysfunction (e.g. the inability to achieve and sustain an erection).

ELIGIBILITY:
Inclusion Criteria:

* Males >18 years of age suffering from sexual dysfunction

Exclusion Criteria:

* Individuals who have had a prostatectomy - removal of prostate
* Inability to operate the device for any reason
* Females
* Males <18 years of age

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
change in modified International Index of Erectile Dysfunction score | baseline and up to 1 month post-baseline
  score 0 to 30 with higher score meaning better erectile function

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eisenberg, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Healthcare, Stanford Hospital, Stanford, California, United States